CLINICAL TRIAL: NCT05568381
Title: Sleep Disturbance in MCI: A Pilot Study of a Cognitive Behavioural Therapy Digital Intervention (SUCCEED)
Brief Title: Sleep Disturbance in MCI: A Study of a Cognitive Behavioural Therapy Digital Intervention
Acronym: SUCCEED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sydney (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021/761
Record Dates: First submitted 2022-08-23; First posted 2022-10-05 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Cognitive Dysfunction; Insomnia; Mild Cognitive Impairment; Cognitive Disorder; Sleep Wake Disorders
Keywords: Mild cognitive impairment; Insomnia; Cognitive Behavioral Therapy; Aging; Sleep; Digital; Older people
MeSH Terms: conditions — Cognitive Dysfunction; Sleep Initiation and Maintenance Disorders; Sleep Wake Disorders

STUDY DESIGN:
Intervention Model Description: Eligible participants will be randomly allocated (1:1) to the intervention or wait-listed control arm. Participants allocated to the digital CBT-I arm (intervention) will receive the commercially available program. The program provides an online media-rich course of CBT-I delivered by an animated "virtual therapist". This will be available for participants for 12 weeks. A wait-listed control of sleep health education will consist of 3 modules delivered biweekly of generalised sleep health information that could be found on the internet.
Masking Description: This is an open label study as participants will be informed immediately of their allocated group by an automatic email and/or text message (dependent on participant preference). Therefore, participants will not be blind to treatment allocation. Self-report questionnaires and cognitive tests will be completed online
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Digital Cognitive Behavioural therapy for insomnia (Experimental): Participants will receive a commercially available 6-week, online media-rich course of CBT-I delivered by an animated "virtual therapist" (Sleepio). Treatment content of this intervention includes behavioural components (sleep restriction, stimulus control, and relaxation), cognitive components (paradoxical intention, cognitive restructuring, mindfulness, positive imagery, and 'putting the day to rest') and educational components (psychoeducation and sleep hygiene). Each of the 6 sessions lasts ~ 30 minutes and incorporates an initial progress review in relation to individualised goals, and exploration of self-reported diary data relating to the participant's current sleep status and pattern. The full program can be accessed via a website or iOS app. Participants will have access to the intervention for up to 12 weeks.
  Interventions: Device: digital CBT-I
- Sleep Health Education wait-list control (Active Comparator): Those in the control group will have access to three modules of the Sleep Health Education package following completion of baseline questionnaires. Each module will be delivered fortnightly with basic information about sleep health (e.g. the impact of sleep on health, creating a sleep-conducive bedroom, sleep and mood). Participants will receive a link to access each module as they are made available.
  At trial completion (week 12), control participants will be offered the opportunity to engage with digital CBT-I.
  Interventions: Other: Online Sleep Health Education package

INTERVENTIONS:
Device: digital CBT-I — Sleepio is a digital cognitive behavioral therapy (CBT) program designed to treat insomnia. The program is fully automated, and its underlying algorithms drive the delivery of information, support, and advice.
  Other Names: Sleepio
  Arms: Digital Cognitive Behavioural therapy for insomnia
Other: Online Sleep Health Education package — Wait-listed control participants will have full access to three online modules for the duration of the study. The information in these modules will provide non-tailored basic sleep information and content will contain text and basic images but will not be personalised to the individual participant.
  Arms: Sleep Health Education wait-list control

SUMMARY:
This study aims to determine the feasibility of a randomized-controlled trial of digital cognitive behavioural therapy for insomnia (CBT-I) for sleep and cognitive performance in older adults with MCI and insomnia symptoms (50-80 years). The trial will be completed online, and participants will be recruited from the community across Australia.

DETAILED DESCRIPTION:
Insomnia is a highly prevalent sleep disorder which affect approximately 10% of the adult population and 40% of the older population. Further, insomnia has been linked to an increased risk of developing dementia. Currently, the recommended first-line treatment for insomnia is cognitive behavioural therapy for insomnia (CBT-I), in both face-to-face and digital form. Despite the strong evidence for digital CBT-I, there are insufficient data regarding the benefits and effectiveness of digital CBT-I in older people with mild cognitive impairment (MCI).

The investigators will conduct a fully online study comparing 6-weeks of digital behavioural therapy for insomnia (CBT-I) against online sleep health education. Participants will be recruited using social media, as well as from memory clinics. Participants will be screened and determined eligibility and consent will be conducted online. Subsequently, participants will be randomly allocated to either digital CBT-I delivered via an application called Sleepio or wait-listed control. The Sleepio app is a sleep-improvement program that uses cognitive behavioural therapy techniques to improve insomnia symptoms. The wait-listed control will consist of 3 modules of an online Sleep Health Education package delivered fortnightly with non-tailored basic sleep information. They will be directed to a website to determine eligibility and then provided access to either the digital CBT-I (Sleepio) or the wait-listed control with a link to the first online module.

At baseline, all participants will complete self-reported measures of subjective cognitive complaints, insomnia, fatigue, sleep, depression, quality of life, and digital health literacy. Also, they will complete three web-based cognitive assessments that measure memory, processing speed, and executive functioning. These will be repeated at follow-up at weeks 12

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MCI as defined by a neuropsychologist.
* Able to provide informed electronic consent.
* Fluent English literacy.
* Adults aged between 50-80 years.
* Insomnia symptoms as indicated by a score >10 on the Insomnia Severity Index (ISI).
* Regular computer, smartphone, or tablet use, with internet access.

Exclusion Criteria:

* Previous diagnosis of dementia or a score on the brief Montreal Cognitive Assessment of <18.
* Previous major head injury, cerebrovascular events (stroke, TIA), or loss of consciousness ≥ 30 minutes.
* Previous or current neurological disorder diagnosis (e.g. Parkinson's, multiple sclerosis, epilepsy).
* Current illicit substance use or harmful alcohol intake (Alcohol Use Disorders Identification Test Consumption (AUDIT-C) score > 8).
* Current severe major depression diagnosis as defined by a score >20 on the Patient Health Questionnaire (PHQ-9) and/or suicidal ideation (score of >1 on Q9 of the PHQ-9), or severe psychiatric or developmental disorders (e.g. Schizophrenia, bipolar disorder, autism).
* Major sleep disorders (e.g. narcolepsy, severe restless legs syndrome, and rapid eye movement (REM) sleep behaviour disorder)
* Commencement of continuous positive airway pressure therapy, antidepressants, melatonin or engaged in CBT or psychological interventions within the prior 4 weeks.
* Shift workers, recent (within 30-days) transmeridian travel.
* Older adults with a risk of an increase in daytime sleepiness and decreased alertness (e.g. professional drivers or those who operate heavy machinery).
* Any contraindication to sleep deprivation therapy.
* Currently participating in or has participated in a research study of an investigational agent or device within 4 weeks of enrolment.
* Any medication that has been used to assist sleep for three or more nights per week (e.g. benzodiazepines, sedative hypnotics, opioids) or at the discretion of the clinician.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-04-20 (Actual); Primary Completion 2023-08-10 (Actual); Study Completion 2023-11-17 (Actual)

PRIMARY OUTCOMES:
The proportion of participants who are issued a pre-screening number and then are determined to be eligible to be booked for screening. | During Screening
  The aim is to provide feasibility data for a full-scale randomized controlled trial (RCT). We will document the number of participants who are eligible after the screening process.
The proportion of participants who are issued a screening number and then are determined to be eligible for randomisation. | Over a 6-month period of recruitment.
  We will document the number of participants who consent to the study after all inclusion/exclusion criteria are met.
Percentage of participants who randomised who originally came from the memory clinic and percentage that were randomised who originally came from online recruitment. | Month 0
  An aim of this trial is to determine the feasibility of recruiting through memory clinics and/or online advertising. We will document the number of participants who have been recruited through memory clinics or online advertising.

SECONDARY OUTCOMES:
Insomnia symptom severity | baseline and at 12 weeks
  Insomnia symptoms severity will be determined from the Insomnia Severity Index (ISI), a 7-item patient reported outcome measure that probes the severity of current symptoms of insomnia over the past 2 weeks. Each item uses a 5-point Likert scale to capture a rating (0 = no problem; 4 = very severe problem) which add up to: no insomnia (0 - 7); sub-threshold insomnia (8 - 14); moderate insomnia (15 - 21); and severe insomnia (22 - 28). Primary endpoint to test for differences is 12 weeks.
Target detection (A'; the accuracy with which a subject detects targets (the expected range is 0.00 to 1.00)) as assessed by the Rapid Visual Processing (RVP) test from the Cambridge Neuropsychological Test Automatic Battery (CANTAB). | baseline and at 12 weeks
  The RVP is a web-based test from CANTAB that measures sustained attention. The outcome is auto-calculated by CANTAB. Primary endpoint to test for differences is 12 weeks.
Processing speed (median response latency in milliseconds) as assessed by the Rapid Visual Processing (RVP) test from the Cambridge Neuropsychological Test Automatic Battery (CANTAB). | baseline and at 12 weeks
  The RVP is a web-based test from CANTAB that measures sustained attention. The outcome is auto-calculated by CANTAB. Primary endpoint to test for differences is 12 weeks.
Adjusted perseveration (number of times that the subject chose a wrong stimulus adjustment for every stage that was not reached) as assessed by Intra-Extra Dimensional Set Shift (IED) subtest from CANTAB. | baseline and at 12 weeks
  The IED is a web-based test from CANTAB that assess executive functioning. The outcome is auto-calculated by CANTAB. Primary endpoint to test for differences is 12 weeks.
Visual memory (number of times the subject chose the incorrect box for a stimulus adjusted for the estimated number of errors on trials not completed) as assessed by the Paired Associate Learning (PAL) subtest from CANTAB. | baseline and at 12 weeks
  The PAL is a web-based test from CANTAB that assess visual memory and new learning. The outcome is auto-calculated by CANTAB. Primary endpoint to test for differences is 12 weeks.
Problem solving (number of trials completed on all attempted stages with an adjustment for any stages not reached) as assessed by Intra-Extra Dimensional Set Shift (IED) subtest from the Cambridge Neuropsychological Test Automatic Battery (CANTAB). | baseline and at 12 weeks
  The IED is a web-based test from CANTAB that assess executive functioning. The outcome is auto-calculated by CANTAB. Primary endpoint to test for differences is 12 weeks.
Depressive symptoms | baseline and at 12 weeks
  Depressive symptoms will be assessed by the Geriatric Depression Scale (GDS) which is a 15-item self-report questionnaire that has been developed to assess depressive symptoms This instrument evaluated depressive symptoms using yes/no answers. Scores range between 0 and 15 points where higher scores indicate more severe depressive symptoms. Primary endpoint to test for differences is 12 weeks.

OTHER OUTCOMES:
Overall health status | baseline and at 12 weeks
  Overall health status will be assessed using the EuroQol 5-dimension scale, a brief questionnaire about health-related quality of life that queries 5 dimensions of everyday experience that are each rated using a 5-point scale (no problems/slight problems/moderate problems/severe problems/extreme problems) and the overall score range from 0 (worst health state imaginable) to 100 (best health state imaginable). Primary endpoint to test for differences is 12 weeks.
Adherence to the online modules | by 12 weeks
  The digital CBT-I program provides online analytics which can be used to monitor adherence by assessing what proportion of patients in the Sleepio arm complete at least 4 sessions. Thus, adherence to the online modules will be determined using a pre-specified value of ≥4 sessions
Overall engagement to digital CBT-I | by 12 weeks
  Overall engagement to digital CBT-I will be assessed by the User Engagement Scale Short Form (UES-SF). The UES-SF is composed of 12 questions divided between 4 domains: aesthetic appeal (AE), reward (RW), perceived usability (PU) and focused attention (FA). Overall engagement score will be calculated by adding all of the items together and dividing by twelve. The overall score ranges from 1 (low engagement) to 5 (high engagement). This is a tool that has been used to evaluate the main factors for adherence in online interventions.
Self-report sleep quality | baseline and at 12 weeks
  Self-report sleep quality will be determined from the Pittsburgh Sleep Quality Index (PSQI), a 19-items questionnaire with 7 components. Each of these components produces a score ranging from 0 (no difficulty) to 3 (severe difficulty). The components scores are summed to yield a global score (range 0 - 21) with higher total score indicating worse sleep quality. Primary endpoint to test for differences is 12 weeks.
Self-report sleep efficiency | baseline and at 12 weeks
  Self-report sleep efficiency will be determined from the Pittsburgh Sleep Quality Index (PSQI), a 19-items questionnaire with a global score range 0 - 21 with higher total score indicating worse sleep quality. Component 4 of the PSQI will be calculated using the question about sleep duration, bedtime and risetime and analysed as a raw percentage for differences at 12 weeks.
Fatigue levels | baseline and at 12 weeks
  Fatigue levels will be determined from the Flinders Fatigue Scale (FSS), a 7 items self-report scale which assess fatigue over the past 2 weeks. This scale provides a total fatigue score ranging from 0 to 31, with higher scores indicating greater fatigue. Primary endpoint to test for differences is 12 weeks.
Subjective cognitive complaints | baseline and at 12 weeks
  Subjective cognitive complaints will be determined from the British Columbia Cognitive Complaints Inventory, a 6-item screening tool that assesses perceived cognitive difficulties in the past 7 days. Each item uses a 3-point Likert scale to capture a rating (0 = not at all; 3= very much) which add up to: broadly normal (0-4); mild cognitive complaints (5-8); moderate cognitive complaints (9-14); and severe cognitive complaints (15-18). Primary endpoint to test for differences is 12 weeks.
Target detection (number of correct hits) as assessed by the Rapid Visual Processing (RVP) test from the Cambridge Neuropsychological Test Automatic Battery (CANTAB). | baseline and at 12 weeks
  The RVP is a web-based test from CANTAB that measures sustained attention. The outcome is auto-calculated by CANTAB. Primary endpoint to test for differences is 12 weeks.
Probability of False Alarm (False Alarms ÷ (False Alarms + Correct Rejections)) as assessed by the Rapid Visual Processing (RVP) test from the Cambridge Neuropsychological Test Automatic Battery (CANTAB). | baseline and at 12 weeks
  The RVP is a web-based test from CANTAB that measures sustained attention. The outcome is auto-calculated by CANTAB. Primary endpoint to test for differences is 12 weeks.
New learning (number of times a subject chose the correct box on their first attempt when recalling the pattern locations. Calculated across all assessed trials) as assessed by the Paired Associate Learning (PAL) subtest from CANTAB. | baseline and at 12 weeks
  The PAL is a web-based test from CANTAB that assess visual memory and new learning. The outcome is auto-calculated by CANTAB. Primary endpoint to test for differences is 12 weeks.
Problem solving (number of times that the subject chose a wrong stimulus) as assessed by Intra-Extra Dimensional Set Shift (IED) subtest from the Cambridge Neuropsychological Test Automatic Battery (CANTAB). | baseline and at 12 weeks
  The IED is a web-based test from CANTAB that assess executive functioning. The outcome is auto-calculated by CANTAB. Primary endpoint to test for differences is 12 weeks.
Perseveration (number of trials for which the outcome was an incorrect response across all assessed trials) as assessed by Intra-Extra Dimensional Set Shift (IED) subtest from the Cambridge Neuropsychological Test Automatic Battery (CANTAB). | baseline and at 12 weeks
  The IED is a web-based test from CANTAB that assess executive functioning. The outcome is auto-calculated by CANTAB. Primary endpoint to test for differences is 12 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Sharon L Naismith, PhD, Principal Investigator — University of Sydney; Camilla Hoyos, PhD, Principal Investigator — University of Sydney
Locations (1):
- The University of Sydney, Sydney, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: Yes
All de-identified data may be shared upon the Principal Investigator's agreement. Ethics approval will be sought prior to any future use of the data.
Supporting Information: Study Protocol, ICF
Time Frame: The study data will be available following all analyses.
Access Criteria: Contact the Principal Investigator to access the data.

REFERENCES:
- [Background] Livingston G, Huntley J, Sommerlad A, Ames D, Ballard C, Banerjee S, Brayne C, Burns A, Cohen-Mansfield J, Cooper C, Costafreda SG, Dias A, Fox N, Gitlin LN, Howard R, Kales HC, Kivimaki M, Larson EB, Ogunniyi A, Orgeta V, Ritchie K, Rockwood K, Sampson EL, Samus Q, Schneider LS, Selbaek G, Teri L, Mukadam N. Dementia prevention, intervention, and care: 2020 report of the Lancet Commission. Lancet. 2020 Aug 8;396(10248):413-446. doi: 10.1016/S0140-6736(20)30367-6. Epub 2020 Jul 30. No abstract available. PMID 32738937
- [Background] Australia D. Dementia Prevalence Data 2018-2058, Commissioned research undertaken by NATSEM: University of Canberra; 2018
- [Background] Sperling RA, Aisen PS, Beckett LA, Bennett DA, Craft S, Fagan AM, Iwatsubo T, Jack CR Jr, Kaye J, Montine TJ, Park DC, Reiman EM, Rowe CC, Siemers E, Stern Y, Yaffe K, Carrillo MC, Thies B, Morrison-Bogorad M, Wagster MV, Phelps CH. Toward defining the preclinical stages of Alzheimer's disease: recommendations from the National Institute on Aging-Alzheimer's Association workgroups on diagnostic guidelines for Alzheimer's disease. Alzheimers Dement. 2011 May;7(3):280-92. doi: 10.1016/j.jalz.2011.03.003. Epub 2011 Apr 21. PMID 21514248
- [Background] Naismith SL, Lewis SJ, Rogers NL. Sleep-wake changes and cognition in neurodegenerative disease. Prog Brain Res. 2011;190:21-52. doi: 10.1016/B978-0-444-53817-8.00002-5. PMID 21531243
- [Background] McKinnon A, Terpening Z, Hickie IB, Batchelor J, Grunstein R, Lewis SJ, Naismith SL. Prevalence and predictors of poor sleep quality in mild cognitive impairment. J Geriatr Psychiatry Neurol. 2014 Sep;27(3):204-11. doi: 10.1177/0891988714527516. Epub 2014 Mar 31. PMID 24687189
- [Background] Xie L, Kang H, Xu Q, Chen MJ, Liao Y, Thiyagarajan M, O'Donnell J, Christensen DJ, Nicholson C, Iliff JJ, Takano T, Deane R, Nedergaard M. Sleep drives metabolite clearance from the adult brain. Science. 2013 Oct 18;342(6156):373-7. doi: 10.1126/science.1241224. PMID 24136970
- [Background] Zachariae R, Lyby MS, Ritterband LM, O'Toole MS. Efficacy of internet-delivered cognitive-behavioral therapy for insomnia - A systematic review and meta-analysis of randomized controlled trials. Sleep Med Rev. 2016 Dec;30:1-10. doi: 10.1016/j.smrv.2015.10.004. Epub 2015 Oct 24. PMID 26615572
- [Background] Winblad B, Palmer K, Kivipelto M, Jelic V, Fratiglioni L, Wahlund LO, Nordberg A, Backman L, Albert M, Almkvist O, Arai H, Basun H, Blennow K, de Leon M, DeCarli C, Erkinjuntti T, Giacobini E, Graff C, Hardy J, Jack C, Jorm A, Ritchie K, van Duijn C, Visser P, Petersen RC. Mild cognitive impairment--beyond controversies, towards a consensus: report of the International Working Group on Mild Cognitive Impairment. J Intern Med. 2004 Sep;256(3):240-6. doi: 10.1111/j.1365-2796.2004.01380.x. PMID 15324367
- [Background] Hu C, Yu D, Sun X, Zhang M, Wang L, Qin H. The prevalence and progression of mild cognitive impairment among clinic and community populations: a systematic review and meta-analysis. Int Psychogeriatr. 2017 Oct;29(10):1595-1608. doi: 10.1017/S1041610217000473. PMID 28884657
- [Background] Jack CR, Wiste HJ, Botha H, Weigand SD, Therneau TM, Knopman DS, Graff-Radford J, Jones DT, Ferman TJ, Boeve BF, Kantarci K, Lowe VJ, Vemuri P, Mielke MM, Fields JA, Machulda MM, Schwarz CG, Senjem ML, Gunter JL, Petersen RC. The bivariate distribution of amyloid-beta and tau: relationship with established neurocognitive clinical syndromes. Brain. 2019 Oct 1;142(10):3230-3242. doi: 10.1093/brain/awz268. PMID 31501889
- [Background] Gauthier S, Reisberg B, Zaudig M, Petersen RC, Ritchie K, Broich K, Belleville S, Brodaty H, Bennett D, Chertkow H, Cummings JL, de Leon M, Feldman H, Ganguli M, Hampel H, Scheltens P, Tierney MC, Whitehouse P, Winblad B; International Psychogeriatric Association Expert Conference on mild cognitive impairment. Mild cognitive impairment. Lancet. 2006 Apr 15;367(9518):1262-70. doi: 10.1016/S0140-6736(06)68542-5. PMID 16631882
- [Background] Love S, Miners JS. Cerebrovascular disease in ageing and Alzheimer's disease. Acta Neuropathol. 2016 May;131(5):645-58. doi: 10.1007/s00401-015-1522-0. Epub 2015 Dec 28. PMID 26711459
- [Background] Toledo JB, Arnold SE, Raible K, Brettschneider J, Xie SX, Grossman M, Monsell SE, Kukull WA, Trojanowski JQ. Contribution of cerebrovascular disease in autopsy confirmed neurodegenerative disease cases in the National Alzheimer's Coordinating Centre. Brain. 2013 Sep;136(Pt 9):2697-706. doi: 10.1093/brain/awt188. Epub 2013 Jul 10. PMID 23842566
- [Background] Naismith SL, Glozier N, Burke D, Carter PE, Scott E, Hickie IB. Early intervention for cognitive decline: is there a role for multiple medical or behavioural interventions? Early Interv Psychiatry. 2009 Feb;3(1):19-27. doi: 10.1111/j.1751-7893.2008.00102.x. PMID 21352171
- [Background] Andrieu S, Coley N, Lovestone S, Aisen PS, Vellas B. Prevention of sporadic Alzheimer's disease: lessons learned from clinical trials and future directions. Lancet Neurol. 2015 Sep;14(9):926-944. doi: 10.1016/S1474-4422(15)00153-2. Epub 2015 Jul 23. PMID 26213339
- [Background] Diamond K, Mowszowski L, Cockayne N, Norrie L, Paradise M, Hermens DF, Lewis SJ, Hickie IB, Naismith SL. Randomized controlled trial of a healthy brain ageing cognitive training program: effects on memory, mood, and sleep. J Alzheimers Dis. 2015;44(4):1181-91. doi: 10.3233/JAD-142061. PMID 25408218
- [Background] Hill NT, Mowszowski L, Naismith SL, Chadwick VL, Valenzuela M, Lampit A. Computerized Cognitive Training in Older Adults With Mild Cognitive Impairment or Dementia: A Systematic Review and Meta-Analysis. Am J Psychiatry. 2017 Apr 1;174(4):329-340. doi: 10.1176/appi.ajp.2016.16030360. Epub 2016 Nov 14. PMID 27838936
- [Background] Gillis C, Mirzaei F, Potashman M, Ikram MA, Maserejian N. The incidence of mild cognitive impairment: A systematic review and data synthesis. Alzheimers Dement (Amst). 2019 Mar 8;11:248-256. doi: 10.1016/j.dadm.2019.01.004. eCollection 2019 Dec. PMID 30911599
- [Background] Barnett JH, Lewis L, Blackwell AD, Taylor M. Early intervention in Alzheimer's disease: a health economic study of the effects of diagnostic timing. BMC Neurol. 2014 May 7;14:101. doi: 10.1186/1471-2377-14-101. PMID 24885474
- [Background] Walker MP. Sleep, memory and emotion. Prog Brain Res. 2010;185:49-68. doi: 10.1016/B978-0-444-53702-7.00004-X. PMID 21075233
- [Background] Naismith SL, Rogers NL, Hickie IB, Mackenzie J, Norrie LM, Lewis SJ. Sleep well, think well: sleep-wake disturbance in mild cognitive impairment. J Geriatr Psychiatry Neurol. 2010 Jun;23(2):123-30. doi: 10.1177/0891988710363710. Epub 2010 Mar 30. PMID 20354239
- [Background] Mander BA, Rao V, Lu B, Saletin JM, Lindquist JR, Ancoli-Israel S, Jagust W, Walker MP. Prefrontal atrophy, disrupted NREM slow waves and impaired hippocampal-dependent memory in aging. Nat Neurosci. 2013 Mar;16(3):357-64. doi: 10.1038/nn.3324. Epub 2013 Jan 27. PMID 23354332
- [Background] Meerlo P, Mistlberger RE, Jacobs BL, Heller HC, McGinty D. New neurons in the adult brain: the role of sleep and consequences of sleep loss. Sleep Med Rev. 2009 Jun;13(3):187-94. doi: 10.1016/j.smrv.2008.07.004. Epub 2008 Oct 9. PMID 18848476
- [Background] Tononi G, Cirelli C. Sleep and the price of plasticity: from synaptic and cellular homeostasis to memory consolidation and integration. Neuron. 2014 Jan 8;81(1):12-34. doi: 10.1016/j.neuron.2013.12.025. PMID 24411729
- [Background] Shokri-Kojori E, Wang GJ, Wiers CE, Demiral SB, Guo M, Kim SW, Lindgren E, Ramirez V, Zehra A, Freeman C, Miller G, Manza P, Srivastava T, De Santi S, Tomasi D, Benveniste H, Volkow ND. beta-Amyloid accumulation in the human brain after one night of sleep deprivation. Proc Natl Acad Sci U S A. 2018 Apr 24;115(17):4483-4488. doi: 10.1073/pnas.1721694115. Epub 2018 Apr 9. PMID 29632177
- [Background] Ohayon MM. Epidemiology of insomnia: what we know and what we still need to learn. Sleep Med Rev. 2002 Apr;6(2):97-111. doi: 10.1053/smrv.2002.0186. PMID 12531146
- [Background] Wolkove N, Elkholy O, Baltzan M, Palayew M. Sleep and aging: 1. Sleep disorders commonly found in older people. CMAJ. 2007 Apr 24;176(9):1299-304. doi: 10.1503/cmaj.060792. PMID 17452665
- [Background] Morin CM, Jarrin DC. Epidemiology of Insomnia: Prevalence, Course, Risk Factors, and Public Health Burden. Sleep Med Clin. 2022 Jun;17(2):173-191. doi: 10.1016/j.jsmc.2022.03.003. Epub 2022 Apr 23. PMID 35659072
- [Background] Roth T. Insomnia: definition, prevalence, etiology, and consequences. J Clin Sleep Med. 2007 Aug 15;3(5 Suppl):S7-10. No abstract available. PMID 17824495
- [Background] Wardle-Pinkston S, Slavish DC, Taylor DJ. Insomnia and cognitive performance: A systematic review and meta-analysis. Sleep Med Rev. 2019 Dec;48:101205. doi: 10.1016/j.smrv.2019.07.008. Epub 2019 Aug 12. PMID 31522135
- [Background] Sterniczuk R, Theou O, Rusak B, Rockwood K. Sleep disturbance is associated with incident dementia and mortality. Curr Alzheimer Res. 2013 Sep;10(7):767-75. doi: 10.2174/15672050113109990134. PMID 23905991
- [Background] Irwin MR, Vitiello MV. Implications of sleep disturbance and inflammation for Alzheimer's disease dementia. Lancet Neurol. 2019 Mar;18(3):296-306. doi: 10.1016/S1474-4422(18)30450-2. Epub 2019 Jan 17. PMID 30661858
- [Background] Shi L, Chen SJ, Ma MY, Bao YP, Han Y, Wang YM, Shi J, Vitiello MV, Lu L. Sleep disturbances increase the risk of dementia: A systematic review and meta-analysis. Sleep Med Rev. 2018 Aug;40:4-16. doi: 10.1016/j.smrv.2017.06.010. Epub 2017 Jul 6. PMID 28890168
- [Background] de Almondes KM, Costa MV, Malloy-Diniz LF, Diniz BS. Insomnia and risk of dementia in older adults: Systematic review and meta-analysis. J Psychiatr Res. 2016 Jun;77:109-15. doi: 10.1016/j.jpsychires.2016.02.021. Epub 2016 Mar 8. PMID 27017287
- [Background] Naismith SL, Mowszowski L. Sleep disturbance in mild cognitive impairment: a systematic review of recent findings. Curr Opin Psychiatry. 2018 Mar;31(2):153-159. doi: 10.1097/YCO.0000000000000397. PMID 29256922
- [Background] D'Rozario AL, Chapman JL, Phillips CL, Palmer JR, Hoyos CM, Mowszowski L, Duffy SL, Marshall NS, Benca R, Mander B, Grunstein RR, Naismith SL. Objective measurement of sleep in mild cognitive impairment: A systematic review and meta-analysis. Sleep Med Rev. 2020 Aug;52:101308. doi: 10.1016/j.smrv.2020.101308. Epub 2020 Mar 13. PMID 32302775
- [Background] Brown BM, Rainey-Smith SR, Bucks RS, Weinborn M, Martins RN. Exploring the bi-directional relationship between sleep and beta-amyloid. Curr Opin Psychiatry. 2016 Nov;29(6):397-401. doi: 10.1097/YCO.0000000000000285. PMID 27584712
- [Background] Brown BM, Rainey-Smith SR, Villemagne VL, Weinborn M, Bucks RS, Sohrabi HR, Laws SM, Taddei K, Macaulay SL, Ames D, Fowler C, Maruff P, Masters CL, Rowe CC, Martins RN; AIBL Research Group. The Relationship between Sleep Quality and Brain Amyloid Burden. Sleep. 2016 May 1;39(5):1063-8. doi: 10.5665/sleep.5756. PMID 27091528
- [Background] Lucey BP, McCullough A, Landsness EC, Toedebusch CD, McLeland JS, Zaza AM, Fagan AM, McCue L, Xiong C, Morris JC, Benzinger TLS, Holtzman DM. Reduced non-rapid eye movement sleep is associated with tau pathology in early Alzheimer's disease. Sci Transl Med. 2019 Jan 9;11(474):eaau6550. doi: 10.1126/scitranslmed.aau6550. PMID 30626715
- [Background] Cross NE, Lagopoulos J, Duffy SL, Cockayne NL, Hickie IB, Lewis SJ, Naismith SL. Sleep quality in healthy older people: relationship with (1)H magnetic resonance spectroscopy markers of glial and neuronal integrity. Behav Neurosci. 2013 Oct;127(5):803-10. doi: 10.1037/a0034154. PMID 24128367
- [Background] Elcombe EL, Lagopoulos J, Duffy SL, Lewis SJ, Norrie L, Hickie IB, Naismith SL. Hippocampal volume in older adults at risk of cognitive decline: the role of sleep, vascular risk, and depression. J Alzheimers Dis. 2015;44(4):1279-90. doi: 10.3233/JAD-142016. PMID 25408219
- [Background] McKinnon AC, Lagopoulos J, Terpening Z, Grunstein R, Hickie IB, Batchelor J, Lewis SJ, Duffy S, Shine JM, Naismith SL. Sleep disturbance in mild cognitive impairment is associated with alterations in the brain's default mode network. Behav Neurosci. 2016 Jun;130(3):305-15. doi: 10.1037/bne0000137. Epub 2016 Mar 10. PMID 26963234
- [Background] Brett J, Murnion B. Management of benzodiazepine misuse and dependence. Aust Prescr. 2015 Oct;38(5):152-5. doi: 10.18773/austprescr.2015.055. Epub 2015 Oct 1. PMID 26648651
- [Background] Lovato N, Lack L, Wright H, Kennaway DJ. Evaluation of a brief treatment program of cognitive behavior therapy for insomnia in older adults. Sleep. 2014 Jan 1;37(1):117-26. doi: 10.5665/sleep.3320. PMID 24470701
- [Background] Naismith SL, Pye J, Terpening Z, Lewis S, Bartlett D. "Sleep Well, Think Well" Group Program for Mild Cognitive Impairment: A Randomized Controlled Pilot Study. Behav Sleep Med. 2019 Nov-Dec;17(6):778-789. doi: 10.1080/15402002.2018.1518223. Epub 2018 Sep 24. PMID 30247939
- [Background] Cassidy-Eagle E, Siebern A, Unti L, Glassman J, O'Hara R. Neuropsychological Functioning in Older Adults with Mild Cognitive Impairment and Insomnia Randomized to CBT-I or Control Group. Clin Gerontol. 2018 Mar-Apr;41(2):136-144. doi: 10.1080/07317115.2017.1384777. Epub 2017 Dec 8. PMID 29220627
- [Background] Miller, C. B., Espie, C. A., & Kyle, S. D. (2014). Cognitive behavioral therapy for the management of poor sleep in insomnia disorder. ChronoPhysiology and Therapy, 4, 99.
- [Background] Freeman D, Sheaves B, Goodwin GM, Yu LM, Nickless A, Harrison PJ, Emsley R, Luik AI, Foster RG, Wadekar V, Hinds C, Gumley A, Jones R, Lightman S, Jones S, Bentall R, Kinderman P, Rowse G, Brugha T, Blagrove M, Gregory AM, Fleming L, Walklet E, Glazebrook C, Davies EB, Hollis C, Haddock G, John B, Coulson M, Fowler D, Pugh K, Cape J, Moseley P, Brown G, Hughes C, Obonsawin M, Coker S, Watkins E, Schwannauer M, MacMahon K, Siriwardena AN, Espie CA. The effects of improving sleep on mental health (OASIS): a randomised controlled trial with mediation analysis. Lancet Psychiatry. 2017 Oct;4(10):749-758. doi: 10.1016/S2215-0366(17)30328-0. Epub 2017 Sep 6. PMID 28888927
- [Background] Pillai V, Anderson JR, Cheng P, Bazan L, Bostock S, Espie CA, Roth T, Drake CL. The Anxiolytic Effects of Cognitive Behavior Therapy for Insomnia: Preliminary Results from a Web-delivered Protocol. J Sleep Med Disord. 2015;2(2):1017. Epub 2015 Feb 23. PMID 32195356
- [Background] Kyle SD, Hurry MED, Emsley R, Marsden A, Omlin X, Juss A, Spiegelhalder K, Bisdounis L, Luik AI, Espie CA, Sexton CE. The effects of digital cognitive behavioral therapy for insomnia on cognitive function: a randomized controlled trial. Sleep. 2020 Sep 14;43(9):zsaa034. doi: 10.1093/sleep/zsaa034. PMID 32128593
- [Background] Cheng P, Luik AI, Fellman-Couture C, Peterson E, Joseph CLM, Tallent G, Tran KM, Ahmedani BK, Roehrs T, Roth T, Drake CL. Efficacy of digital CBT for insomnia to reduce depression across demographic groups: a randomized trial. Psychol Med. 2019 Feb;49(3):491-500. doi: 10.1017/S0033291718001113. Epub 2018 May 24. PMID 29792241
- [Background] Luik AI, Bostock S, Chisnall L, Kyle SD, Lidbetter N, Baldwin N, Espie CA. Treating Depression and Anxiety with Digital Cognitive Behavioural Therapy for Insomnia: A Real World NHS Evaluation Using Standardized Outcome Measures. Behav Cogn Psychother. 2017 Jan;45(1):91-96. doi: 10.1017/S1352465816000369. Epub 2016 Jul 26. PMID 27456542
- [Background] Cuamatzi-Castelan, A. S., Cheng, P., Fellman-Couture, C., Tallent, G., Tran, K. M., Espie, C. A., ... & Drake, C. L. (2018). 0375 Long-term Efficacy of the Sleep to Prevent Evolving Affective Disorders (SPREAD) Trial as an Internet-based Treatment for Insomnia. Sleep, 41, A143
- [Background] LaMonica HM, English A, Hickie IB, Ip J, Ireland C, West S, Shaw T, Mowszowski L, Glozier N, Duffy S, Gibson AA, Naismith SL. Examining Internet and eHealth Practices and Preferences: Survey Study of Australian Older Adults With Subjective Memory Complaints, Mild Cognitive Impairment, or Dementia. J Med Internet Res. 2017 Oct 25;19(10):e358. doi: 10.2196/jmir.7981. PMID 29070481
- [Background] Bastien CH, Vallieres A, Morin CM. Validation of the Insomnia Severity Index as an outcome measure for insomnia research. Sleep Med. 2001 Jul;2(4):297-307. doi: 10.1016/s1389-9457(00)00065-4. PMID 11438246
- [Background] LaMonica HM, Davenport TA, Roberts AE, Hickie IB. Understanding Technology Preferences and Requirements for Health Information Technologies Designed to Improve and Maintain the Mental Health and Well-Being of Older Adults: Participatory Design Study. JMIR Aging. 2021 Jan 6;4(1):e21461. doi: 10.2196/21461. PMID 33404509
- [Background] Manea L, Gilbody S, McMillan D. Optimal cut-off score for diagnosing depression with the Patient Health Questionnaire (PHQ-9): a meta-analysis. CMAJ. 2012 Feb 21;184(3):E191-6. doi: 10.1503/cmaj.110829. Epub 2011 Dec 19. PMID 22184363
- [Background] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Background] Rey, A. (1941). L'examen psychologique dans les cas d'encéphalopathie traumatique.(Les problems.). Archives de psychologie.
- [Background] Wechsler D. Wechsler Memory Scale. San Antonio (TX): Psychological Corporation; 1997
- [Background] Lezak MD, Howieson DB, Loring DW, Fischer JS. Neuropsychological assessment. Oxford University Press, USA; 2004.
- [Background] Wechsler D. Wechsler Adult Intelligence Scale-Fourth Edition: Technical and interpretative manual. San Antonio (TX): Pearson Assessment; 2008.
- [Background] Roth C. (2011) Boston Naming Test. In: Kreutzer J.S., DeLuca J., Caplan B. (eds) Encyclopedia of Clinical Neuropsychology. Springer, New York, NY. https://doi.org/10.1007/978-0-387-79948-3_869
- [Background] Smith A. Symbol digit modalities test: Manual. Los Angeles (CA): Western Psychological Services; 1982.
- [Background] Ricker JH, Axelrod BN. Analysis of an Oral Paradigm for the Trail Making Test. Assessment. 1994 Mar;1(1):47-52. doi: 10.1177/1073191194001001007. PMID 9463499
- [Background] Petersen RC, Doody R, Kurz A, Mohs RC, Morris JC, Rabins PV, Ritchie K, Rossor M, Thal L, Winblad B. Current concepts in mild cognitive impairment. Arch Neurol. 2001 Dec;58(12):1985-92. doi: 10.1001/archneur.58.12.1985. PMID 11735772
- [Background] Busse A, Hensel A, Guhne U, Angermeyer MC, Riedel-Heller SG. Mild cognitive impairment: long-term course of four clinical subtypes. Neurology. 2006 Dec 26;67(12):2176-85. doi: 10.1212/01.wnl.0000249117.23318.e1. PMID 17190940
- [Background] Chung F, Yegneswaran B, Liao P, Chung SA, Vairavanathan S, Islam S, Khajehdehi A, Shapiro CM. STOP questionnaire: a tool to screen patients for obstructive sleep apnea. Anesthesiology. 2008 May;108(5):812-21. doi: 10.1097/ALN.0b013e31816d83e4. PMID 18431116
- [Background] Norman CD, Skinner HA. eHEALS: The eHealth Literacy Scale. J Med Internet Res. 2006 Nov 14;8(4):e27. doi: 10.2196/jmir.8.4.e27. PMID 17213046
- [Background] Cameron K, Williamson P, Short MA, Gradisar M. Validation of the Flinders Fatigue Scale as a measure of daytime fatigue. Sleep Med. 2017 Feb;30:105-112. doi: 10.1016/j.sleep.2016.11.016. Epub 2016 Dec 3. PMID 28215232
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Sheikh, J. I., & Yesavage, J. A. (1986). Geriatric Depression Scale (GDS): recent evidence and development of a shorter version. Clinical Gerontologist: The Journal of Aging and Mental Health.
- [Background] Iverson GL, Lam RW. Rapid screening for perceived cognitive impairment in major depressive disorder. Ann Clin Psychiatry. 2013 May;25(2):135-40. PMID 23638444
- [Background] Espie CA, Kyle SD, Miller CB, Ong J, Hames P, Fleming L. Attribution, cognition and psychopathology in persistent insomnia disorder: outcome and mediation analysis from a randomized placebo-controlled trial of online cognitive behavioural therapy. Sleep Med. 2014 Aug;15(8):913-7. doi: 10.1016/j.sleep.2014.03.001. Epub 2014 Mar 12. PMID 24791643
- [Background] Espie CA, Kyle SD, Williams C, Ong JC, Douglas NJ, Hames P, Brown JS. A randomized, placebo-controlled trial of online cognitive behavioral therapy for chronic insomnia disorder delivered via an automated media-rich web application. Sleep. 2012 Jun 1;35(6):769-81. doi: 10.5665/sleep.1872. PMID 22654196
- [Background] Miller CB, Espie CA, Epstein DR, Friedman L, Morin CM, Pigeon WR, Spielman AJ, Kyle SD. The evidence base of sleep restriction therapy for treating insomnia disorder. Sleep Med Rev. 2014 Oct;18(5):415-24. doi: 10.1016/j.smrv.2014.01.006. Epub 2014 Feb 12. PMID 24629826
- [Background] Kyle SD, Morgan K, Spiegelhalder K, Espie CA. No pain, no gain: an exploratory within-subjects mixed-methods evaluation of the patient experience of sleep restriction therapy (SRT) for insomnia. Sleep Med. 2011 Sep;12(8):735-47. doi: 10.1016/j.sleep.2011.03.016. Epub 2011 Sep 9. PMID 21907616